CLINICAL TRIAL: NCT02374645
Title: A Phase Ib, Open-label, Multi-centre Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-tumour Activity of Volitinib in Combination With Gefitinib in Patients With Epidermal Growth Factor Receptor-mutated Non-small Cell Lung Cancer Who Have Progressed on Epidermal Growth Factor Receptor Inhibitor Treatment
Brief Title: A Phase I Study of Safety and Pharmacokinetics of Volitinib in Combination With Gefitinib in EGFR(+) NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5080C00001
Record Dates: First submitted 2015-02-12; First posted 2015-03-02 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Volitinib (AZD6094) 600mg + gefitinib 250 mg (Experimental): Cohort 1: Volitinib（AZD6094） 600 mg od + gefitinib 250 mg od
  Interventions: Drug: Volitinib; Drug: gefitinib
- Volitinib (AZD6094) 800mg + gefitinib 250 mg (Experimental): Cohort 2: Volitinib（AZD6094） 800 mg od + gefitinib 250 mg od
  Interventions: Drug: gefitinib

INTERVENTIONS:
Drug: Volitinib — 600mg or 800mg QD: Patients may continue to receive the treatment as long as they are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: AZD6094; HMPL-504
  Arms: Volitinib (AZD6094) 600mg + gefitinib 250 mg
Drug: gefitinib — 250mg QD: Patients may continue to receive the treatment as long as they are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: Iressa; ZD1839

SUMMARY:
This is a Phase 1b, open-label, multicentre study of AZD6094 in combination with gefitinib in patients with epidermal growth factor receptor (EGFR) mutation positive (m+) and progressed on EGFR Tyrosine kinase inhibitor (TKI) treatment.

DETAILED DESCRIPTION:
A total of 53 patients will be enrolled in the safety run-in and expansion phases:

* Safety run-in phase - patients with EGFR mutation-positive (EGFRm+), locally advanced or metastatic non-small cell lung cancer (NSCLC), who have progressed on previous EGFT TKI treatment.In the safety run-in phase of the study, the sample size may vary, depending on the number of dose levels evaluated and the number of Dose Limiting Toxicities (DLTs) observed in each cohort.
* Expansion phase - patients who are EGFRm+ and cMet-positive with locally advanced or metastatic NSCLC, who have progressed on previous EGFR-TKI treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures. If a patient declines to participate in any voluntary exploratory research and/or genetic component of the study there will be no penalty or loss of benefit to the patient and he or she will not be excluded from other aspects of the study.
2. Male or female aged at least 18 years and older.
3. Histologically or cytologically confirmed locally advanced or metastatic NSCLC patients who are harbouring an EGFR mutation known to be associated with EGFR-TKI sensitivity (including exon 19 deletion, L858R, L861Q, G719X). Local test for EGFR mutation is acceptable. In the expansion phase, patients must have a positive cMet test by a central laboratory. Safety run-in phase: EGFR mutation positive. A local EGFR test result is acceptable Expansion phase: EGFR mutation positive and cMet-positive. cMet test is performed by a central lab.
4. Radiological documentation of disease progression while on a previous continuous treatment with EGFR-TKI eg, gefitinib or erlotinib. All patients must have documented radiological progression on the last treatment administered prior to enrolling in the study. The patients must have been treated with an EGFR-TKI with objective clinical benefit (CR/PR) or SD for 3 months, and who have subsequently shown radiological progression on treatment. In addition, other lines of therapy may have been given.
5. At least 1 lesion, not previously irradiated, not biopsied during the screening period, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) which is suitable for accurate repeated measurements.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks.
7. Women should agree to use adequate contraceptive measures (as defined in section 5.1), should not be breast feeding, and must have a negative pregnancy test prior to start of dosing or if of child-bearing potential or of non-child- bearing potential must have evidence of this by fulfilling 1 of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments
   * Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation
   * Women under 50 years of age would be considered postmenopausal if they have been amenorrhoeic for at least 12 months following the cessation of exogenous hormonal treatments, and have serum follicle-stimulating hormone (FSH) and luteinizing hormone (LH) levels in the postmenopausal range for the institution.
8. Sexually active male patients should be willing to use barrier contraception; ie, condoms.
9. For inclusion in the genetic research, patients must provide informed consent for genetic research.

Exclusion Criteria:

1. Intervention with any of the following:

   * Treatment with an EGFR-TKI within approximately 5x half-life (eg, within 8 days for erlotinib, gefitinib or afatanib, within 10 days for dacomitinib) of the first dose of study treatment
   * Any cytotoxic chemotherapy, investigational agents or other anticancer drugs for the treatment of advanced NSCLC from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment
   * Patients currently receiving (or unable to stop use at least 2 weeks) prior to receiving the first dose of AZD6094, medications known to be strong inhibitors of CYP1A2 (Appendix E)
   * Prior or current treatment with AZD6094 or another cMet inhibitor (eg, foretinib, crizotinib, cabozantinib, onartuzumab)
   * Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable.
2. Radiotherapy with a limited field of radiation for palliation within 1 week of the first dose of study treatment, with the exception of patients receiving radiation to more than 30% of the bone marrow or with a wide field of radiation which must be completed ≥4 weeks of the first dose of study treatment.
3. Major surgical procedure, (excluding placement of vascular access) or significant traumatic injury within 4 weeks of the first dose of study treatment, or have an anticipated need for major surgery during the study
4. With the exception of alopecia and CTCAE Grade 2, prior chemotherapy-related neuropathy, any unresolved toxicities from prior therapy and/or pre-study biopsies greater than CTCAE Grade 1 at the time of starting study treatment
5. Have non-measurable disease at baseline per RECIST v1.1. To ensure that the patient will be able to complete the evaluable period of the study and the assessment of progression can be performed according to the RECIST v1.1 criteria and the relevant treatment decisions applied OR can be summarised for patients with measurable disease at baseline
6. Presence of other active cancers, or history of treatment for invasive cancer ≤5 years. Patients with Stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
7. Current leptomeningeal metastases or spinal cord compression. Brain metastases are only permitted if treated, asymptomatic, and stable (not requiring steroids for at least 4 weeks prior to start of study treatment).
8. Patients with known tumour thrombus or deep vein thrombosis are eligible if stable on low molecular weight heparin for ≥4 weeks.
9. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, renal transplant, active bleeding diatheses, which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol; including evidence of active infection including hepatitis B (HBV) surface antigen, hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
10. Any serious uncontrolled medical disorder or active infection that would impair the patient's ability to receive IP, such as conditions associated with frequent diarrhoea.
11. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTc) >470 msec obtained from triplicate ECGs
    * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG; eg, complete left bundle branch block, third degree heart block, second degree heart block, PR interval >250 msec
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalaemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age or any concomitant medication known to prolong the QT interval- Inadequately controlled hypertension (ie, systolic blood pressure (BP) >160 mmHg or diastolic BP >100 mmHg (patients with values above these levels must have their BP controlled with medication prior to starting treatment).
    * Atrial fibrillation with a ventricular rate >100 bpm on ECG at rest
    * Symptomatic heart failure - New York Heart Association (NYHA) Grade II-IV
    * Unstable angina pectoris
    * Acute myocardial infarction
    * Uncontrolled angina (Canadian Cardiovascular Society Grade II-IV despite medical therapy)
    * Stroke or transient ischemic attack in the last 6 months
12. Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

    * Absolute neutrophil count <1.5x109/L
    * Platelet count <100x109/L
    * Haemoglobin <90 g/L
    * Alanine aminotransferase (ALT) >2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
    * Aspartate aminotransferase (AST) >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases
    * Total bilirubin (TBL) >1.5 times ULN, TBL >3 times ULN in patients with documented Gilbert's Syndrome (unconjugated hyperbilirubinaemia) or in the presence of liver metastases
    * Creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation), confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN
13. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD6094 or gefitinib
14. History of hypersensitivity to active or inactive excipients of AZD6094 or gefitinib or drugs with a similar chemical structure or class to AZD6094 or gefitinib. Unable to undergo an MRI or contrast CT procedures
15. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD. Insufficient lung function dependent on supplemental oxygen (determined by either clinical examination or an arterial oxygen tension (PaO2) of <70 Torr)
16. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
17. Involvement in the planning and conduct of the study (applies to AstraZeneca staff or staff at the study site)
18. Previous enrolment in the present study

    In addition, the following are considered criteria for exclusion from the exploratory genetic research:
19. Previous allogeneic bone marrow transplant
20. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-02-18 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Number of adverse events and serious adverse events | From ICF signed to within 28 days after the last dose
  the grade of AE event according to CTC AE 4.0

SECONDARY OUTCOMES:
The Pharmacokinetics (PK) profiles of AZD6094 | Cycle 1 Day1 and Day 15
  Peak Plasma Concentration (Cmax)
The Pharmacokinetics (PK) profiles of AZD6094 | Cycle 1 Day1 and Day 15
  Area under the plasma concentration versus time curve (AUC)
Progression-free survival (PFS） | from enrolled until progression or death due to any cause, assessed up to 2 year
  6-months PFS, 12 months PFS and 24 month PFS
Disease control rate（DCR) | 12 weeks and 24 weeks
  CR+PR+SD

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Prof., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong General Hospital, Guangzhou, China

REFERENCES:
- [Derived] Yang JJ, Fang J, Shu YQ, Chang JH, Chen GY, He JX, Li W, Liu XQ, Yang N, Zhou C, Huang JA, Frigault MM, Hartmaier R, Ahmed GF, Egile C, Morgan S, Verheijen RB, Mellemgaard A, Yang L, Wu YL. A phase Ib study of the highly selective MET-TKI savolitinib plus gefitinib in patients with EGFR-mutated, MET-amplified advanced non-small-cell lung cancer. Invest New Drugs. 2021 Apr;39(2):477-487. doi: 10.1007/s10637-020-01010-4. Epub 2020 Oct 14. PMID 33052556